CLINICAL TRIAL: NCT04392804
Title: Efficacy of Intraseptal Anesthesia Obtained by 4 % Articaine With 1:100,000 Epinephrine Achieved by Computer-controlled Delivery System
Brief Title: Efficacy of Intraseptal Anesthesia of 4% Articaine With Epinephrine Achieved by Computer-controlled Delivery System
Acronym: EISAAECCLAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Natasa Nikolic Jakoba, Associate professor, DDS, MSc, PhD, University of Belgrade
Other Study IDs: UBelgrade 36/8
Record Dates: First submitted 2020-05-09; First posted 2020-05-19 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia, Local; Periodontitis
Keywords: intraseptal anesthesia; ISA; CCLADS
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 0.1 ml 4% articaine: single dose of 0.1 ml 4% articaine with 1:100,000 epinephrine delivered by computer-controlled local delivery system (Anaject), in purpose for scaling and root planing
  Interventions: Procedure: scaling and root planing
- 0.2 ml 4% articaine: single dose of 0.2 ml 4% articaine with 1:100,000 epinephrine delivered by computer-controlled local delivery system (Anaject), in purpose for scaling and root planing
  Interventions: Procedure: scaling and root planing
- 0.3 ml 4% articaine: single dose of 0.3 ml 4% articaine with 1:100,000 epinephrine delivered by computer-controlled local delivery system (Anaject), in purpose for scaling and root planing
  Interventions: Procedure: scaling and root planing

INTERVENTIONS:
Procedure: scaling and root planing — one appointment for scaling and root planing of selected periodontal pockets, with periodontal curette (HuFriedy, Chicago, IL, USA), rinsing with saline solution

SUMMARY:
The aims of our study were to evaluate the clinical anesthetic parameters of the intraseptal anesthesia (ISA), achieved by computer-controlled local anesthetic delivery system CCLADS, for scaling and root planing, as a primary outcome of the study. In addition, as secondary outcome of the study the impact of destruction of the periodontal supporting tissues on clinical anesthetic parameters of the ISA achieved by 4% articaine with 1:100,000 epinephrine, using CCLAD system.

DETAILED DESCRIPTION:
After including the patients into the study, patient needs to sign a written consent. After that, the next appointment will be scheduled. On the next appointment, each patient included in this study will undergo ultrasound cleaning and receive guidance for adequate everyday oral hygiene. The next appointment, after 10 days will be scaling and root planing for selected periodontal pockets. Because it is painful treatment, anesthesia is needed to be administrated. Patients will be split into three groups by picking cards, for receiving different doses of 4% articaine with 1:100,000 epinephrine ORABLOC® (40 mg/ml Articaine + 0.01 mg/ml Epinephrine, PIERREL S.P.A, Capua, Italy) in each group. Doses will be 0.1 ml, 0.2 ml, and 0.3 ml of 4% articaine with epinephrine for one appointment scaling and root planing. Anesthesia will be obtained by CCLADS device Anaject® (Septodont, Sallanches, Franc). The Intraseptal anesthesia (ISA) will be the method of administrating the anesthesia. Parameters of the device will be a mode with constant pressure, injection speed - mode LOW 0.005 ml/s. Time for application will depend on the dose, and it will be 20 s for 0.1 ml, 40 s for 0.2 ml, and 60 s for 0.3 ml.

Parameters of local anesthesia will be recorded by the pin-prick test. The pain will be rated by the visual-analogue scale (VAS). The pain will be rated immediately upon termination of the local anesthetic delivery and during the scaling and root planing.

Patients will be followed up the next day for local side effects and their need for analgesic medication.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* confirmed diagnosis of periodontitis
* presence of minimum 20 teeth
* absence of decay
* preserved tooth vitality
* good systematic health

Exclusion Criteria:

* allergy to articaine with 1: 100,000 epinephrine
* pregnancy
* lactation
* medication uptake that affects the periodontal supporting tissues
* acute pain, swelling, presence of gingival lesions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy periodontitis patients having the indication for scaling and root planing.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of success anesthesia | 1 day
  The number of success anesthesia
Duration of soft tissue anesthesia | 1 day
  Time from completion of the injection until patient start filling discomfort/pain on pinprick test, measured in minutes.
Width of the anesthetic field | 1 day
  Distance between two needles that were not causing pain on pinprick test, measured in millimeters.
Onset time for anesthesia | 1 day
  Time started after completion of the injection until profound anesthesia is establish, measured in seconds.
Rate of pain during anesthetic delivery by VAS | 1 day
  Visual analogue scale (VAS) is a scale graded from 0 to 100 mm, where 0 is labeled for the minimum feel of pain or no pain, and 100 is labeled for maximum feel of pain (unbearable pain). Patient is placing a mark on the horizontal scale depending on the intensity of the pain sensation.
Rate of pain during scaling and root planing by VAS | 1 day
  Visual analogue scale (VAS) is a scale graded from 0 to 100 mm, where 0 is score for the minimum feel of pain or no pain, and 100 is score for maximum feel of pain (unbearable pain). Patient is placing a mark on the horizontal scale depending on the intensity of the pain sensation.
Presence of side effects | 1 day
  Record any side effects.
Analgesic medication consumption | 1 day
  Record number of analgesic medications.
Wich day analgesic medication is used | 7 days
  Wich day from intervention a analgesic medication is used

SECONDARY OUTCOMES:
Pocket probing depths | 1 day
  Measuring the pocket probing depths by periodontal probe, in milimeteres.
Gingival margin level | 1 day
  Measuring the gingival margin level by periodontal probe, in milimeteres.
Clinical attachment level | 1 day
  Measuring the clinical attachment level by periodontal probe, measured in milimeters.
Percentage of bleeding sites | 1 day
  The number of sites where bleeding is recorded is divided by the total number of available sites in the mouth and multiplied by 100 to express the bleeding index as a percentage.
Percentage of plaque index | 1 day
  The number of sites where plaque is recorded is divided by the total number of available sites in the mouth and multiplied by 100 to express the plaque index as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Oral medicine, School of Dental Medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
no, for now, need to review conditions of terms of sharing the information

REFERENCES:
- [Derived] Djoric J, Djinic Krasavcevic A, Barac M, Kuzmanovic Pficer J, Brkovic B, Nikolic-Jakoba N. Patient discomfort and intensity of intraseptal anesthesia of computer-controlled articaine/epinephrine delivery for scaling and root planing. Clin Oral Investig. 2023 Oct;27(10):6221-6234. doi: 10.1007/s00784-023-05238-1. Epub 2023 Aug 29. PMID 37644233
- [Derived] Djoric J, Djinic Krasavcevic A, Barac M, Kuzmanovic Pficer J, Brkovic B, Nikolic-Jakoba N. Efficacy of intraseptal anesthesia obtained by computer-controlled articaine with epinephrine delivery in scaling and root planing. Clin Oral Investig. 2023 Jun;27(6):2913-2922. doi: 10.1007/s00784-023-04889-4. Epub 2023 Feb 6. PMID 36746819